CLINICAL TRIAL: NCT04878939
Title: Evaluation of Incisors' Position Following Anterior Segment Retraction Using Friction Versus Frictionless Mechanics: A Randomized Clinical Trial
Brief Title: Evaluation of Incisors' Position Following Anterior Segment Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Dorra Bakhit, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FUE.REC 11/10-2018
Record Dates: First submitted 2021-04-25; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Bimaxillary Protrusion
Keywords: friction; frictionless; CBCT; anterior segment retraction; T loop

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the main investigator to the interventions was difficult, yet the outcome assessor was masked to the intervention and assessed unidentified CBCTs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior segment retraction using sliding mechanics (friction) (Experimental): Power chain
  Interventions: Other: Power chain used for anterior segment retraction
- Anterior segment retraction using segmental mechanics (frictionless) (Experimental): T-loop
  Interventions: Other: T-loop fabricated to perform anterior segment retraction

INTERVENTIONS:
Other: Power chain used for anterior segment retraction — Elastomeric chain rendering 160 g/side extending between mini-screw implant and a hook crimped on 0.017- by 0.025-inch stainless steel wire distal to the lateral incisor.
  Arms: Anterior segment retraction using sliding mechanics (friction)
Other: T-loop fabricated to perform anterior segment retraction — In the frictionless group, anterior segment retraction was done using closing T-loops fabricated from 0.017- by 0.025-inch titanium molybdenum alloy (TMA) wire rendering comparable retraction force.
  Arms: Anterior segment retraction using segmental mechanics (frictionless)

SUMMARY:
There's scarcity in literature concerning the issue of anterior segment retraction technique and its effect on anterior teeth position. Therefore, a randomized clinical trial has been chosen to investigate this issue, aiming to support clinicians with the best guidelines for anterior segment retraction.

DETAILED DESCRIPTION:
Thirty females with bimaxillary protrusion were randomly allocated into two groups. In one group, anterior segment retraction was commenced using an elastomeric chain rendering 160 g/side extending between mini-screw implant and a hook crimped on 0.017- by 0.025-inch stainless steel wire distal to the lateral incisor. In the other group, anterior segment retraction was done using closing T-loops fabricated from 0.017- by 0.025-inch titanium molybdenum alloy (TMA) wire rendering comparable retraction force. Three-dimensional analysis of incisors' buccolingual (BL)- torque, mesiodistal (MD)- tip, vertical position changes and root resorption were assessed using cone beam computed tomography scans.

ELIGIBILITY:
Inclusion Criteria:

* Female patients (Age 13- 25 y)
* Class I molar relation (Angle's classification)
* Bimaxillary protrusion requiring extraction of four first premolars and maximum anchorage.
* full permanent dentition (except 3rd molars)
* Good general and oral health

Exclusion Criteria:

* Systemic disease or syndromes or on anti-inflammatory medication.
* Extracted or missing permanent teeth (other than 3rd molars)
* Badly decayed teeth (other than 1st premolars)
* Parafunctional habits
* History of previous orthodontics treatment

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Torque of the incisors | through study completion (Pre/post retraction), an average of 6 months
  The change of the outer angle between long axis of each upper anterior tooth and palatal plane on CBCT pre and post retracation and the change in the outer angle between long axis of each lower anterior tooth and horizontal plane on CBCT pre and post retracation
Tip of the incisors | through study completion (Pre/post retraction), an average of 6 months
  The change of the angle between the long axis of the incisors and mid-sagittal plane on CBCT pre and post retracation
Vertical changes of the incisors | through study completion (Pre/post retraction) , an average of 6 months
  The change of the linear distance between the centroid of each maxillary anterior tooth and palatal Plane on CBCT pre and post retracation and The change of the linear distance between centroid of each mandibular anterior tooth and horizontal Plane on CBCT pre and post retracation

SECONDARY OUTCOMES:
Root resorption of the anterior teeth | through study completion (Pre/post retraction), an average of 6 months
  measuring the amount of resorption using CBCT in mm pre and post retraction

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, Professor and Chairman, Study Director — Future University in Egypt
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be ready to share after publication

REFERENCES:
- [Derived] Bakhit DMI, Tawfik MGY, Dehis HM, Mostafa YA, El Sharaby FA. Position and root resorption of the incisors following anterior segment retraction using friction versus frictionless mechanics: A randomised controlled trial. J Orthod. 2025 Mar;52(1):12-21. doi: 10.1177/14653125241261402. Epub 2024 Jul 25. PMID 39049618

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04878939/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04878939/ICF_001.pdf